CLINICAL TRIAL: NCT01323296
Title: Ferumoxytol for Magnetic Resonance Imaging of Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 10/S1103/50 (REC REF)
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2010-10

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Magnetic resonance; Nanoparticle; Iron; Inflammation
MeSH Terms: conditions — Myocardial Infarction; Inflammation | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferumoxytol (Active Comparator): Patients will be administered intravenous ferumoxytol 1 - 3 days following myocardial infarction after baseline cardiac magnetic resonance scanning.
  Interventions: Other: Ferumoxytol
- Control (No Intervention): Subjects who have suffered myocardial infarction will undergo cardiac magnetic resonance imaging at the same time points as those in the 'ferumoxytol' arm but will not receive ferumoxytol or placebo.

INTERVENTIONS:
Other: Ferumoxytol — One dose of intravenous ferumoxytol (4 mgFe/kg body weight at a rate of up to 1 mL/sec)
  Other Names: Feraheme; Advanced Magnetics, Inc., Cambridge, MA
  Arms: Ferumoxytol

SUMMARY:
The investigators wish to examine whether a novel 'nanoparticle' of iron oxide, administered intravenously allows an area of heart muscle damage after heart attack to be visualised using a magnetic resonance scanner.

DETAILED DESCRIPTION:
Using ferumoxtran (Feraheme) as a USPIO contrast agent for magnetic resonance imaging at 3 Tesla, we aim to conduct the first clinical study to examine the utility of this novel contrast agent to image myocardial inflammation after myocardial infarction.

We will test the following hypotheses in patients who have suffered recent acute myocardial infarction.

1. Intravenous injection of ferumoxytol accumulates at the site of myocardial infarction and this can be visualised by magnetic resonance imaging.
2. The spatial extent of the MRI signal change evoked by ferumoxytol in the myocardium is proportional to the volume of infarcted myocardium (as assessed by a gadolinium late-enhancement study).
3. Myocardial MRI signal change evoked by ferumoxytol is positively correlated with blood markers of systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Presentation with myocardial infarction (either 'ST-elevation' myocardial infarction or 'non-ST-elevation' myocardial infarction
* Troponin I ≥ 10 IU/mL at 12 hours after the onset of chest pain
* Age 18 - 80 years inclusive

Exclusion Criteria:

* Known critical (≥95%) left main stem coronary artery disease
* Continued symptoms of angina at rest or minimal exertion
* Atrial fibrillation
* Symptomatic heart failure; Killip Class ≥2.
* Hepatic failure (Childs-Pugh grade B or C) or renal failure (estimated glomerular filtration rate <25 mL/min)
* Contraindication to magnetic resonance imaging
* Past history of systemic iron overload/haemochromatosis
* Patients with known allergy to dextran- or iron-containing compounds

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in myocardial T2* magnetic resonance signal | Before, 1 day, 2 days, 4 days, 1 week and 1 month post ferumoxytol
  Change in T2*weighted myocardial signal as assessed by magnetic resonance imaging before and after ferumoxytol administration.

SECONDARY OUTCOMES:
Change in systemic blood markers of inflammation | Before, 1 day, 2 days, 4 days, 1 week and 1 month after administration of ferumoxytol
  Change in systemic (blood) markers of inflammation over time after myocardial infarction and correlation with T2*weighted MR signal after administration of ferumoxytol.

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, FRCP, PhD, Principal Investigator — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - Royal Infirmary of Edinburgh, Edinburgh, Midlothian
  - University of Edinburgh, Edinburgh, Midlothian

REFERENCES:
- [Derived] Alam SR, Shah AS, Richards J, Lang NN, Barnes G, Joshi N, MacGillivray T, McKillop G, Mirsadraee S, Payne J, Fox KA, Henriksen P, Newby DE, Semple SI. Ultrasmall superparamagnetic particles of iron oxide in patients with acute myocardial infarction: early clinical experience. Circ Cardiovasc Imaging. 2012 Sep 1;5(5):559-65. doi: 10.1161/CIRCIMAGING.112.974907. Epub 2012 Aug 8. PMID 22875883